CLINICAL TRIAL: NCT00380172
Title: A Multicenter, Open Label, Prospective Study to Determine Safety and Efficacy Over an Additional 12-Month Period With Non-Exudative Age-Related Macular Degeneration (With Follow-on to 12-Months)
Brief Title: Long-Term Efficacy in AMD of Rheopheresis in North America
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: OccuLogix (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMD-03-02
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2006-09-25 (Estimated); Status verified 2006-09

CONDITIONS: Macular Degeneration
Keywords: AMD; Macular Degeneration; Retinal Degeneration
MeSH Terms: conditions — Macular Degeneration; Retinal Degeneration

INTERVENTIONS:
Device: Rheopheresis blood filtration

SUMMARY:
The purpose of these studies are to evaluate the effect on vision in subjects with AMD who received active and placebo treatment in the MIRA-1 study.

ELIGIBILITY:
Inclusion Criteria:

* Must have participated in treatment arm of MIRA-1 trial and completed 4 treatments and 6 and 9 month follow up visits.
* Dry AMD in at least one eye.
* Available for study duration of 12 months.
* Weigh >110 lbs.
* If on lipid-lowering medication must remain on for duration of trial. If not, must agree to not initate during trial.
* Normal Pt/ PTT. If on coumadin, at the discretion of the investigator.
* Must be highly motivated, alert and oriented, and able to provide consent.
* Agree to discontinue current ocular vitamin regimen and take uniform supplement provided by the sponsor.

Exclusion Criteria:

* Both eyes wet AMD.
* Condition limiting view of the fundus.
* Poor general health or unstable diseases.
* HCT < 35%, evidence of active bleeding, platelet count <100000 K/uL, prolonged Pt/ PTT, or significant coagupapathies.
* significant cardiac problems.
* Uncontrolled hypertension.
* History of CVA of TIA within a year.
* Significant hepatic, renal, or pulmonary disease, or insulin dependent diabetes.
* Allergy to fluorescein sodium and indocyanine green (ICG), heparin, ACDA, local anesthetics, or adhesive tape.
* Pregnant or breastfeeding women, or women of childbearing potential not using chemical or mechanical contraception.
* Investigation trial within 30 days.
* Major surgery within 30 days.
* Unwilling to adhere to visit schedule.
* Unstable medical of psychological condition.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2005-10; Study Completion 2007-10

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the change from baseline and ETDRS visual acuity in subjects with non-exudative AMD who participated in AMD-02-99.

SECONDARY OUTCOMES:
The secondary objective of this study is to evaluate the safety of rheopheresis filtration treatments in subjects with non-exudative AMD as measured by AE's early DC's and Lab evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Nozhat Choudry', Ph.D., Study Director — OccuLogix, Inc.
Locations (9):
- United States (8):
  - Retina Vitreous Associates, Beverly Hills, California
  - Aran Eye Associates, Coral Gables, Florida
  - Retina Health Care, Fort Myers, Florida
  - The Macula Center, Palm Harbor, Florida
  - UIC Eye Center, Chicago, Illinois
  - Macula Care, New York, New York
  - Carolina Eye Associates, Southern Pines, North Carolina
  - Associated Retinal Consultants, Bala-Cynwyd, Pennsylvania
- W. Bradley Kates, MD, Oakville, Ontario, Canada